CLINICAL TRIAL: NCT06623370
Title: The Effect of Methylprednisolone Administration on the Reversal Time of Rocuronium by Sugammadex in the Pediatric Patient Group
Brief Title: The Effect of Methylprednisolone on the Reversal Time of Rocuronium by Sugammadex in the Pediatric Patient Group
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, MUSTAFA BÜYÜKCAVLAK, Medical Doctor, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 34028104-799
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Sugammadex Reversal Time; Muscle Weakness
Keywords: sugammadex; methylprednisolone; reversal time; rocuronium; pediatric patients
MeSH Terms: conditions — Muscle Weakness | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Active Comparator): In addition to the routine anesthesia protocol, 1 mg/kg of methylprednisolone will be administered after induction.
  Interventions: Drug: methylprednisolone
- Group C (Placebo Comparator): Routine anesthesia will be administered.
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: methylprednisolone — Patients will undergo standard noninvasive blood pressure monitoring, electrocardiogram, peripheral oxygen saturation (SpO2), and capnography. After anesthesia induction, neuromuscular monitoring will also be applied. Anesthesia induction will be performed with 2-4 mg/kg propofol and 1 mcg/kg fentanyl. First group (Group M), patients will receive 1 mg/kg methylprednisolone , while in the second group (Group C), patients will receive 5 ml of normal saline. Immediately afterward, the neuromuscular monitor will be set to measure the Train of Four (TOF). Following this, 0.6-1.2 mg/kg of rocuronium will be administered intravenously. If necessary, additional doses of 0.15 mg/kg rocuronium will be given during the operation when TOF count reaches T2. For postoperative analgesia, 15 mg/kg of i.v. paracetamol will be administered. At the end of the surgery, when anesthesia is terminated and T2 reappears in TOF count, all patients will receive a single bolus injection of sugammadex.
  Arms: Group M
Other: Saline (NaCl 0,9 %) (placebo) — Patients will undergo standard noninvasive blood pressure monitoring, electrocardiogram, peripheral oxygen saturation (SpO2), and capnography. After anesthesia induction, neuromuscular monitoring will also be applied. Anesthesia induction will be performed with 2-4 mg/kg propofol and 1 mcg/kg fentanyl. First group (Group M), patients will receive 1 mg/kg methylprednisolone , while in the second group (Group C), patients will receive 5 ml of normal saline. Immediately afterward, the neuromuscular monitor will be set to measure the Train of Four (TOF). Following this, 0.6-1.2 mg/kg of rocuronium will be administered intravenously. If necessary, additional doses of 0.15 mg/kg rocuronium will be given during the operation when TOF count reaches T2. For postoperative analgesia, 15 mg/kg of i.v. paracetamol will be administered. At the end of the surgery, when anesthesia is terminated and T2 reappears in TOF count, all patients will receive a single bolus injection of sugammadex.
  Arms: Group C

SUMMARY:
The aim of this study is to thoroughly investigate the interaction between methylprednisolone and sugammadex in the pediatric patient population. Our hypothesis is that methylprednisolone will interact with sugammadex, leading to a prolonged reversal time of rocuronium by sugammadex and, at the same time, a reduction in the effect profile of methylprednisolone.

Approximately 80 volunteers will be included in the study. Patients will not have any additional responsibilities related to this study. There are no risks or benefits to patients associated with this research. The study will begin immediately before the patient's surgery and will end two hours after the operation. Volunteers participating in the study will be randomly assigned to one of two groups: one group will receive methylprednisolone during surgery, and the other group will not. Methylprednisolone is a medication used to prevent postoperative pain, swelling, nausea, and vomiting. If these complaints are detected in patients from either group after surgery, appropriate treatments will be administered to alleviate them.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to provide informed consent and reliably report symptoms to the research team,
* Classified as Physical Status 1 and 2 according to the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* Patients for whom parental or personal consent could not be obtained
* ASA Physical Status 3 or higher
* Known history of allergic reactions to the drugs specified in the protocol
* Patients requiring emergency surgery
* Expected difficult airway
* Preoperative corticosteroid use
* Presence of respiratory system diseases
* Presence of neuromuscular diseases
* Presence of enzymatic or endocrine disorders
* Presence of liver or kidney failure
* Presence of cardiovascular diseases
* Patients with abnormal cognitive or physical development
* History of treatment with drugs that have a high potential for interaction with sugammadex (e.g., toremifene, flucloxacillin, fusidic acid).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
reversal time | The study will conclude after the patient has been postoperatively monitored for 2 hours in the recovery unit
  The time to reach a TOF ratio of 0.9 after sugammadex administration and the time until extubation will be recorded for all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buyukcavlak M, Tire Y, Mermer A, Yuce MS, Yildirim SN, Kozanhan B. The effect of methylprednisolone on the reversal time of rocuronium by sugammadex in the paediatric patient group: A randomised controlled trial. Eur J Anaesthesiol. 2025 Nov 1;42(11):1025-1033. doi: 10.1097/EJA.0000000000002241. Epub 2025 Jul 16. PMID 40673736